CLINICAL TRIAL: NCT04433234
Title: A Phase II, Long-term, Extension Study of DS-5141b in Patients With Duchenne Muscular Dystrophy
Brief Title: Long-term, Extension Study of DS-5141b in Patients With Duchenne Muscular Dystrophy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS5141-A-J201; 205321 (Other: JapicCTI)
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; DMD; Oligonucleotides, antisense; Exon skipping; DS-5141b
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DS-5141b 2.0 mg/kg (Experimental): Participants who will receive DS-5141b 2.0 mg/kg once weekly.
  Interventions: Drug: DS-5141b
- DS-5141b 6.0 mg/kg (Experimental): Participants who will receive DS-5141b 6.0 mg/kg once weekly.
  Interventions: Drug: DS-5141b

INTERVENTIONS:
Drug: DS-5141b — Administered via subcutaneous injection once weekly
  Other Names: Renadirsen

SUMMARY:
This is a multicenter, open-label, long-term, extension, phase 2 study to evaluate the safety and efficacy of long-term treatment with DS-5141b in patients with DMD who have completed DS5141-A-J101.

ELIGIBILITY:
Inclusion Criteria:

* Has competed a study of DS5141-A-J101

Exclusion Criteria:

* Significant safety issues in a study of DS5141-A-J101
* Patient who does not consent to use appropriate contraception
* Patient not appropriate to participant in the study as determined by the Investigator

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 8 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | From first injection to after the last injection of DS-5141b in this study (within approximately 2 years)
Change in distance walked during 6-minute walk test (6MWT) | Every 3 months (within approximately 2 years)
Change in time to stand (TTSTAND) | Every 3 months (within approximately 2 years)
Change in time in Timed up and go test | Every 3 months (within approximately 2 years)
Change in time in 10-meter Run/Walk test | Every 3 months (within approximately 2 years)
Change in score in the North Star Ambulatory Assessment (NSAA) | Every 3 months (within approximately 2 years)
Change in score in the Performance of Upper Limb (PUL) | Every 3 months (within approximately 2 years)
Change in Left Ventricular Ejection Fraction percentage (LVEF %) | Every 6 months (within approximately 2 years)
Change in in Forced Vital Capacity (FVC) (percent predicted) | Every 6 months (within approximately 2 years)
Change in Muscle Strength Measured by Quantitative Muscle Strength Assessment | Every 3 months (within approximately 2 years)

SECONDARY OUTCOMES:
Concentration of DS-5141a in plasma | Every 3 months (within approximately 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo Co., Ltd.
Locations (2):
- Japan (2):
  - National Center of Neurology and Psychiatry, Tokyo, Kodaira-Shi
  - Kobe University Hospital, Hyōgo

IPD SHARING:
Plan to Share IPD: No